CLINICAL TRIAL: NCT05146856
Title: Impact of a Modified Schedule Including a Day Without Clinical Activity Before Night Shift on Non-technical Skills of French Residents in Intensive Care Unit, a Prospective Randomized Multi Center Study: REPOPREGARD Protocol Study
Brief Title: Impact of a Day Without Clinical Activity Before Night Shift on Non-technical Skills of Intensive Care Residents
Acronym: REPOPREGARD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2021 LAUTRETTE REPOPREGARDE
Record Dates: First submitted 2021-10-18; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-10

CONDITIONS: Physician Fatigue
Keywords: Personnel Staffing and Scheduling; High fidelity simulation; Medical Errors / prevention & control; Psychomotor Performance / physiology; Sleep; Work Schedule Tolerance; Internship and Residency / organization & administration; Cross-Over Studies; Humans

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Residents in control group have a usual day with clinical activity before night shift
- Intervention: Residents in intervention group have a day off clinic before night shift (i.e day off or day with university activity)

SUMMARY:
In this proposal, investigators seek to address conclusively two knowledge gaps: 1) the lack of data on the impact of a schedule including a day off clinic before night shift on performances of residents in anesthesia or critical care medicine and 2) the lack of data on the relationship between resident sleep deprivation and their non technical skills impairment. Investigators designed a prospective, randomized, blinded in cross over evaluation of medical pratices. Investigators will compare resident's performance during a high fidelity simulation session, on crisis managment in intensive care unit, after a night shift in intensive care unit, of residents who work on an intervention schedule with no clinical activity before night shift, with resident's performance of residents who had a traditionnal schedule including an usual clinical day before night shift. Investigators also assess cognitive performances, sleepiness and self esteem before and after night shift. Investigators specific aims will be:

To test the hypothesis that residents working on an intervention schedule will have non technical skills, assessed by Ottawa GRS global score, significantly less impaired after a night shift, than those on traditionnal schedule

To test the hypothesis that residents working on an interveniton schedule will have cognitive performances, sleepiness and self esteem less impaired after night shift than those on a traditionnal schedule

DETAILED DESCRIPTION:
Main objective of this study is to compare the non-technical skills after night shift, of anaesthesia and critical care residents who did not have clinical activity before the night shift with those who had at least 8 hours of clinical activity before. The workforce is constrained by the number of residents in training at Clermont-Ferrand and Lyon University Public Hospital. Thus, it is possible to consider the inclusion of 60 residents for 55 evaluable. With such numbers, the clinically relevant difference of 6 points for the Ottawa GRS score (for a standard deviation of 11) can be demonstrated with an alpha risk of bilateral error of 5% and a power of 80%. Two interim analyzes will be carried out including the first 20 interns and then 20 additional interns (therefore for 40 interns) with the aim of stopping the study for "effectiveness", more precisely stopping the study for evidence of a statistically significant difference for the primary outcome measure, with risks of first error observed respectively at 0.0005 and 0.014 comparisons (correction due to multiples). A simulation of the statistical power will also be proposed during the performance of these analyzes; if necessary, a new estimation of the workforce will be proposed to the competent authorities. Investigators do not plan loss of follow up.

ELIGIBILITY:
Inclusion Criteria:

* residents in Anesthesia or Critical care medicine
* Who effect night shift in intensive care unit
* Able to take a day off clinic before night shift
* Able to give consent

Exclusion Criteria:

* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will include volunteer residents in anesthesia of critical care medicine of Gabriel Montpied university hospital of Clermont Ferrand.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Residents' non technical skills after a night shift | Immediatly after the end of the night shift
  Measured by Ottawa Global Rated Scale global score assessed during a high fidelity simulation session of crisis managment. Global score is comprise between 7 for a performance expected from a beginner and 42 for a performance expeted from an expert.

SECONDARY OUTCOMES:
Residents' non technical skill before a night shift | Baseline, before the night shift
  Measured by Ottawa Global Rated Scale global score assessed during a high fidelity simulation session of crisis managment. Global score is comprise between 7 for a performance expected from a beginner and 42 for a performance expeted from an expert.
Cognitive performances : Phasic alert test | Before the night shift
  refers to the notion of general wakefulness allowing to react quickly and appropriately to requests, score obtained from computer tool
Cognitive performances : Phasic alert test | After the night shift up to 12 hours
  refers to the notion of general wakefulness allowing to react quickly and appropriately to requests, score obtained from computer tool
Cognitive performances : Divided attention test | Before the night shift
  refers to the notion of paying attention to several things at the same time, score obtained from computer tool
Cognitive performances : Divided attention test | After the night shift up to 12 hours
  refers to the notion of paying attention to several things at the same time, score obtained from computer tool
Cognitive performances : Flexibility test with alternation | Before the night shift
  refers to the notion of displacement of the attentional focus, score obtained from computer tool
Cognitive performances : Flexibility test with alternation | After the night shift up to 12 hours
  refers to the notion of displacement of the attentional focus, score obtained from computer tool
Cognitive performances : Working memory test | Before the night shift
  refers to the notion of maintaining and updating when carrying out complex problems, score obtained from computer tool
Cognitive performances : Working memory test | After the night shift up to 12 hours
  refers to the notion of maintaining and updating when carrying out complex problems, score obtained from computer tool
Cognitive performances : Computerized Speed Cognitive Test | Before the night shift
  refers to the notion of the speed of information processing, score obtained from computer tool
Cognitive performances : Computerized Speed Cognitive Test | After the night shift up to 12 hours
  refers to the notion of the speed of information processing, score obtained from computer tool
Sleepiness | Before the night shift
  Measured by Karolinska Sleepiness scale, a score of 1 for a great tiredness to 9 for a very well awake state.
Sleepiness | After the night shift up to 12 hours
  Measured by Karolinska Sleepiness scale, a score of 1 for a great tiredness to 9 for a very well awake state.
Self esteem | Before the night shift
  Measured by Rosenberg Self Esteem scale, a score lower than 25 indicates a low self esteem and a score higher than 39 indicates a high self esteem.
Self esteem | After the night shift up to 12 hours
  Measured by Rosenberg Self Esteem scale, a score lower than 25 indicates a low self esteem and a score higher than 39 indicates a high self esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No